CLINICAL TRIAL: NCT00856050
Title: Phase 2 Clinical Study of Letrozole in Women With Advanced Estrogen/Progesterone Receptor Positive Uterine Leiomyosarcoma
Brief Title: Letrozole in Women With Advanced Estrogen/Progesterone Receptor Positive Uterine Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Suzanne George, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-341
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Leiomyosarcoma
Keywords: estrogen receptor positive; progesterone receptor positive; letrozole
MeSH Terms: conditions — Leiomyosarcoma | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- letrozole (Experimental): single arm trial - all patients received letrozole 2.5mg by mouth per day
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — Taken orally once a day continuously
  Other Names: Femara

SUMMARY:
The purpose of this research study is to determine if letrozole is effective at controlling the growth or spread of estrogen and/or progesterone receptor positive uterine leiomyosarcoma. This drug has been used in research studies for other cancers and is currently approved by the FDA for use in breast cancer. Because letrozole lowers hormone levels in the body, it may be helpful to control tumors that express hormone receptors ( ER/PR).

DETAILED DESCRIPTION:
* Participants will take letrozole orally once a day. During the research study the following tests and procedures will be performed:
* Visit 1 (Day 1): physical examination, vital signs and blood work
* Visit 2 (Day 43): physical examination, vital signs, blood work, CT or MRI scan
* Visit 3 (Day 85): physical examination, vital signs, blood work, CT or MRI scan
* Participants will remain on the study drug as long as they do not have any serious sife effect and their disease does not get worse

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, advanced estrogen (ER)/progesterone receptor (PR) positive leiomyosarcoma of uterine origin, for which standard multi-modality curative therapies do not exist or are no longer effective
* Patients must be postmenopausal. Postmenopausal is defined as any of the following: 1)Bilateral oophorectomy 2) 60 years of age or older 3)Younger than 60 AND amenorrheic for 12 months or more AND follicle stimulating hormone (FSH) and estradiol (E2) within postmenopausal range 4)Ovarian ablation radiotherapy confirmed by FSH and estradiol (E2) level in the postmenopausal range
* Evidence of ER and/or PR positivity, either in primary or secondary tumor tissue
* Measurable disease outside of a prior irradiated area as defined by RECIST guidelines. A lesion in a previously irradiated area is not eligible for measurable diseae unless there is objective evidence of progression of the lesion prior to study enrollment
* 18 years of age or older
* Life expectancy of 3 months or more
* ECOG Performance Status 0, 1, or 2
* No limit to number of prior chemotherapies or biologics
* Normal organ function as outlined in the protocol
* Resolution of clinically significant toxicities related to prior therapies

Exclusion Criteria:

* Pre-menopausal women
* Participants who have had systemic anti-cancer therapy within 3 weeks of study entry (8 weeks for nitrosoureas or mitomycin C)
* Palliative radiotherapy within 2 weeks of study entry
* Major surgery within 2 weeks of study entry
* Prior hormonal therapy for the treatment of uterine leiomyosarcoma (prior hormone replacement therapy is allowed)
* Participants may not be receiving any other concomitant investigational agents
* Uncontrolled brain or central nervous system metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to letrozole
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Individuals with a history of a different malignancy, other than cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy OR other primary malignancy is neither currently clinically significant nor requiring active intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 patients were enrolled, and 26 patients received at least one dose of study medication and were included in the analysis.
Groups:
- Letrozole: Experimental: letrozole single arm trial - all patients received letrozole 2.5mg by mouth per day
Period: Overall Study
Arm/Group | Letrozole
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 27 patients were enrolled, and 26 patients received at least one dose of study medication and were included in the analysis.
Groups:
- Letrozole: letrozole 2.5mg by mouth per day
Arm/Group | Letrozole
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 56 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 12 Weeks
Description: Data below are reported as progression free rate (%).
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Letrozole
Number analyzed (Participants) | 26
percentage of participants | 46 [29 to 64]

ADVERSE EVENTS:
Arm/Group | Letrozole
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 20/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Letrozole (N=26)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2/25
Nausea (Gastrointestinal disorders) | 4/25
Fatigue (General disorders) | 4/25
Joint= pain (Musculoskeletal and connective tissue disorders) | 5/25
Muscle= pain (Musculoskeletal and connective tissue disorders) | 7/25
Hot flashes (Vascular disorders) | 17/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes